CLINICAL TRIAL: NCT00525811
Title: Development of a Web-Based Interactive Patient Decision Aid for the Treatment of Acute Low Back Pain and Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Prof. Dr. Dr. Martin Haerter, University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TK-2005-0111
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Last update posted 2008-06-24 (Estimated); Status verified 2008-06

CONDITIONS: Acute Low Back Pain; Depression
MeSH Terms: conditions — Depression | interventions — Confidentiality

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Interactive decision aid
  Interventions: Other: patient dialogue
- B (Active Comparator): Regular patient information
  Interventions: Other: patient information

INTERVENTIONS:
Other: patient dialogue — Information on shared decision making, how to participate in medical decision making, information on acute low back pain, information on depression
  Arms: A
Other: patient information — Information on acute low back pain, information on depression
  Arms: B

SUMMARY:
Shared decision making (SDM) has been advocated as an appropriate approach for physician patient communication. Positive effects of SDM are e.g higher patient satisfaction, greater treatment adherence, lower decisional conflict and better clinical outcomes. The Section of Clinical Epidemiology and Health Services Research at the University Medical Center in Freiburg (Germany) is developing and evaluating a web-based interactive decision aid ("patient dialogue") to support shared decision making in cooperation with the Techniker Krankenkasse, a large German health insurance company. Both development and evaluation are conducted along the International Patient Decision Aid Standards (IPDAS).

The decision aid contains information on acute low back pain and depression and addresses insurance members who are facing a treatment decision in one of the indications. It aims at the development of patient competencies for participating in decision making, the support of constructive health behavior and patients' acceptance of evidence based treatment options.

In an RCT the decision aid will be compared to a regular patient information on a sample of N=500 patients in each group. Data collection will take place at three points of time: before and after use of the decision aid as well as 3 months later.

ELIGIBILITY:
Inclusion Criteria:

* insurance members with acute low back pain or depression

Exclusion Criteria:

* insurance members without symptoms, with chronic back pain, with a bipolar disorder, relatives of people with symptoms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 741 (Actual)
Dates: Start 2007-06; Primary Completion 2008-02 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Decisional conflict | After using the decision aid

SECONDARY OUTCOMES:
Knowledge, Preparation for decision making, Preference for participation, Involvement in decision making, Decision regret, Treatment adherence | After using the decision aid and 3 months later respectively

CONTACTS AND LOCATIONS:
Overall Officials: Martin Haerter, MD, PhD, Study Chair — University Medical Center, Freiburg, Germany
Locations (1):
- University Medical Center, Freiburg im Breisgau, Germany

REFERENCES:
- See also: Related Info — http://www.shared-decision-making.org